CLINICAL TRIAL: NCT01337999
Title: Human Epididymis Protein 4 in Normal Menstruating Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Beth Plante, Beth Plante, M.D., Women and Infants Hospital of Rhode Island
Other Study IDs: 10-0127
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Premenopausal Women
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HE-4 levels, healthy premenopausal women
  Interventions: Other: blood draws

INTERVENTIONS:
Other: blood draws — 5 blood draws during ovulatory menstrual cycles in premenopausal women

SUMMARY:
The purpose of this study is to determine if Human Epididymis Protein 4 (HE-4) levels vary during the menstrual cycles in ovulatory women. HE-4 is a sensitive serological marker that is elevated in certain ovarian and endometrial cancers and can aid in the diagnosis of these malignant conditions. In order to optimize the utility of HE4 as a tumor marker in premenopausal women, its expression in the normal menstrual cycle needs to be characterized. We hypothesize that HE-4 levels do not vary in the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* women age 18-45 years old
* regular menstrual cycles (every 25-35 days)
* normal BMI (19-25)
* no hormonal contraception in the two menstrual cycles prior to enrollment

Exclusion Criteria:

* pregnancy
* pelvic mass

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ovulating women recruited from local college campuses, doctor's offices and hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
HE-4 level | 5 times during menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Beth Plante, M.D., Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Division of Reproductive Endocrinology & Infertility, Providence, Rhode Island, United States

REFERENCES:
- [Background] Anastasi E, Granato T, Marchei GG, Viggiani V, Colaprisca B, Comploj S, Reale MG, Frati L, Midulla C. Ovarian tumor marker HE4 is differently expressed during the phases of the menstrual cycle in healthy young women. Tumour Biol. 2010 Oct;31(5):411-5. doi: 10.1007/s13277-010-0049-1. Epub 2010 May 20. PMID 20490961
- [Background] Moore RG, McMeekin DS, Brown AK, DiSilvestro P, Miller MC, Allard WJ, Gajewski W, Kurman R, Bast RC Jr, Skates SJ. A novel multiple marker bioassay utilizing HE4 and CA125 for the prediction of ovarian cancer in patients with a pelvic mass. Gynecol Oncol. 2009 Jan;112(1):40-6. doi: 10.1016/j.ygyno.2008.08.031. Epub 2008 Oct 12. PMID 18851871
- [Derived] Lambert-Messerlian G, Plante B, Eklund EE, Raker C, Moore RG. Levels of antimullerian hormone in serum during the normal menstrual cycle. Fertil Steril. 2016 Jan;105(1):208-13.e1. doi: 10.1016/j.fertnstert.2015.09.033. Epub 2015 Oct 23. PMID 26477497